CLINICAL TRIAL: NCT04899765
Title: Specific and Non-specific Effects of Measles and BCG Vaccines for Mother and Child
Brief Title: Measles and BCG Vaccines for Mother and Child
Acronym: MATVAC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: The University of Western Australia (Other); Université Libre de Bruxelles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: MATVAC
Record Dates: First submitted 2021-05-18; First posted 2021-05-24 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Vaccine Preventable Disease; Measles; Mother-Infant Interaction; BCG Vaccination Reaction
Keywords: Non-specific effects of vaccines
MeSH Terms: conditions — Vaccine-Preventable Diseases; Measles | interventions — BCG Vaccine; Measles Vaccine

STUDY DESIGN:
Intervention Model Description: We plan a trail randomising non-pregnant women of fertile age 1:1:1 to MV, BCG or placebo. The first children to be born will also be randomised to early MV or no early MV at 20 weeks of age. All children will get the recommended MV by 9 months of age.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: BCG is given intradermally and typically results in a local skin reaction that heals leaving a small scar. Measles vaccine is given subcutaneously and typically does not leave any sign of vaccination. Though we do not believe women will be able to distinguish between intradermal and subcutaneous injections, complete blinding on the recipient side will not be possible; those who get a skin reaction after BCG will most likely be able to guess what they received, whereas MV and placebo recipients will not. We do not believe this will influence the results of the blood testing or their treatment of their offspring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Measles vaccine (Experimental): Measles vaccine in standard dose of 0.5 ml.
  Interventions: Biological: Measles vaccine
- BCG vaccine (Experimental): BCG vaccine in standard dose of 0.1 ml.
  Interventions: Biological: BCG vaccine
- Placebo (Placebo Comparator): Saline injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BCG vaccine — It is an attenuated live bacterial vaccine. This vaccine is a freeze-dried product that must be reconstituted.
  Arms: BCG vaccine
Biological: Measles vaccine — It is an attenuated live virus vaccine. This vaccine is a freeze-dried product that must be reconstituted.
  Arms: Measles vaccine
Other: Placebo — Saline
  Arms: Placebo

SUMMARY:
In Africa, the mortality from infectious diseases remains high. The investigators have discovered that live vaccines such as the BCG vaccine against tuberculosis and the measles vaccine can strengthen resistance to other infections: they have beneficial "non-specific effects". The investigators have now seen signs that these non-specific effects for children are stronger if their mother has been given the same vaccines.

In Africa, BCG vaccine is recommended at birth and measles vaccine at 9 months of age. They are not used beyond childhood.

The investigators will randomize 2400 women to BCG vaccine, measles vaccine, or placebo. The investigators will further randomize their children to an extra early measles vaccine or placebo. The investigators will assess which of the resulting six vaccination schedules are best for women's and children's protection against measles, for the child's immune system, and for general health.

The project will be the first in the world to investigate the importance of vaccinating women with live vaccines.

DETAILED DESCRIPTION:
OBJECTIVES The investigators aim to study the effects of providing measles vaccine (MV) or Bacille Calmette-Guérin vaccine (BCG) to women of fertile age, prior to pregnancy, and to study the added effect of providing MV earlier to their children, for measles-specific and non-specific immunity in the child and for overall health in mother and child.

Specific objectives

To study the interaction of maternal MV and BCG and early infant MV with respect to:

* the magnitude of the measles-specific antibody response in women and children
* the proportion of children with maternal measles antibodies at the time of measles immunization
* the viral load following YF vaccination in children
* overall health in women and children

HYPOTHESES

* Providing MV to women in the fertile age will increase the proportion of children, who are vaccinated in the presence of maternal measles antibody, both at 20 weeks and 9 months of age
* Providing MV or BCG to women in the fertile age will reduce the child's viral load after a YF vaccine provided at 9 months of age
* Providing MV or BCG to women in the fertile age will reduce maternal and child infectious disease morbidity by 20%

METHODS The study will take place at the Bandim Health Project (BHP), Bissau, Guinea-Bissau.

The investigators plan a 3-by-2 factorial trial with randomization of non-pregnant women of fertile age to MV, BCG or placebo, and randomization of their offspring (who will all get BCG at birth according to recommendations) to early MV or no early MV at 20 weeks of age. All children will get the recommended MV by 9 months of age.

The study will enroll 2400 non-pregnant HIV-negative women, who will be randomized 1:1:1 to one of three injections: BCG, MV, or placebo (saline). The first 100 children born to mothers from each of the three groups and surviving until 20 weeks of age will be selected for follow-up. Within strata of maternal vaccination (BCG, MV, placebo) they will be randomized 1:1 to early MV at 20 weeks, or placebo (saline). Thus, a total of 6 groups (A-F) will be formed.

By 9 months of age, 20 children in each randomization group will receive a yellow fever (YF) vaccine and then MV 5 days later. All other children will receive an MV and a YF vaccine when they reach 9 months of age.

Setting:

BHP's Health and Demographic Surveillance System (HDSS) covers six districts in the capital of Guinea-Bissau with around 100,000 individuals. The BHP follows all women of fertile age with monthly visits to register new pregnancies. All children are followed with 4-monthly home visits for infections, hospitalizations, and vaccinations. All vaccinations administered at the three health centers in the study area are documented by BHP. Furthermore, BHP monitors all consultations and admissions at the health centers and all pediatric consultations and admissions at the national hospital.

Enrolment and randomization of women:

Eligible women will be identified through the BHP HDSS. They will receive a home visit by a project assistant, who will explain the study. If they are interested in participating, they will be asked to come to a nearby health center. Here, following informed oral and written consent, a blood sample will be drawn and tested for HIV. If the HIV-test is positive, immediate counseling will be given by a trained project nurse and the woman will be referred to the HIV clinic, per current standard of care. A urine pregnancy test will be carried out. Provided negative HIV and pregnancy tests, an interview regarding background factors, including previous vaccinations, will be carried out. Finally, the woman will be randomized and treated according to the allocation.

Follow-up for pregnancies and morbidity:

Women will be followed for pregnancy. All participating women will also be followed with respect to morbidity (consultations, hospitalizations) at 2-monthly interviews and continuous documentation of hospitalizations and consultations.

Maternal blood samples:

All blood will be collected into Na-Heparin tubes. Baseline blood sample: All women enrolled will have a blood sample obtained by venipuncture at baseline, in conjunction with the HIV screening, just before randomization.

Baseline+4weeks blood sample: A blood sample will be obtained after 4 weeks from 30 women from each group. These samples with be paired with the baseline sample to assess measles-specific antibodies level.

Children:

All children will be followed closely through monthly home visits, during which the mother will be encouraged to bring her child for the scheduled vaccines. At 20 weeks of age, the children will be invited for further randomization.

Inclusion criteria: The first 100 children surviving until 20 weeks of age from each group of enrolled mothers, and having received all recommended vaccines, the 3rd pentavalent vaccine at least 6 weeks before, are eligible for further study randomization.

Exclusion criteria: Exclusion criteria are lack of receipt of all scheduled vaccines, pentavalent vaccine less than 6 weeks ago (in which case children are asked to come back once 6 weeks are reached), and overt illness (in which case they will be referred for treatment and invited to come back when the child is well again).

Randomization of children:

Eligible children are identified at the monthly home visits and asked to come to a nearby health center in the afternoon. Here, provided maternal consent, they will be randomly allocated to early MV or placebo (saline).

Child blood samples:

All blood will be collected into Na-Heparin tubes. Measles specific arm: N=30 from each of Groups A-F: A 2 ml blood sample will be obtained at baseline (either 20 weeks of age or 9 months of age) and a second sample of 2 ml will be obtained at either 9 months of age (those bled first at 20 weeks of age) or 18 weeks after 9-month-vaccination (those bled first at 9 months of age) for assessment of measles-specific antibodies levels.

Non-specific effect arm: N=20 from each of Groups A-F: Children will receive YF vaccine at 9 months of age, a blood sample will be obtained just before and a second sample will be obtained 5 days later for assessment of YF viraemia.

Follow up for child morbidity and mortality:

The 300 children enrolled in the child-vaccination part of the study as well as other children born to the 2400 women enrolled in the maternal vaccination study will be followed for morbidity and mortality. The data collection with be based on the HDSS regular home visits, the registration of consultations in the study area, and the registration of admissions to the pediatric ward of the national hospital.

Vaccination and blinding:

Women vaccination: Women will be vaccinated in right upper arm. The vaccine administrator will know what is given, but the women will not be told before the trial has come to an end.

Child vaccination: MV and YF vaccine will be given subcutaneously according to the national recommendations. Placebo for MV at 20 weeks will be saline, provided subcutaneously in the same volume as MV.

Analysis of blood samples:

The blood samples will be analyzed in collaboration with our international colleagues.

Measles antibodies: Total and measles-specific immunoglobulin G (IgG) levels will be analyzed.

YF vaccine response: Children will receive a single dose of YF vaccine. A blood sample will be obtained 5 days after and tested for yellow fever viral load.

Statistical analysis and sample size:

Maternal and child morbidity data will be analyzed in standard survival analysis for time-to-event data to compare potential differential effects by vaccination allocation. The analysis will take into account other possible interventions or events, campaigns or epidemics, occurring during the period of follow-up.

The study sample size of 2400 women is based on the anticipated delivery rates in the area. Based on census data from BHP, the annual incidence of new deliveries in women with one child of 12 months will be around 15%. Hence, with a cohort of 2,400 enrolled women, it is expected to register >300 deliveries in the 5th -10th trimester after enrolment starts.

ELIGIBILITY:
Inclusion Criteria:

* Female women in the fertile age
* Non-pregnant
* HIV-negative
* Living in the BHP HDSS study area
* Delivered a child that has reached 12 months of age
* Currently not using contraceptives.

Exclusion Criteria:

* Positive pregnancy test
* Positive HIV test
* Tuberculosis (previous or current)
* Immunodeficiency
* Cancer within the last 2 years
* Mid-upper-arm-circumference<200
* Acute ongoing infection

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2400 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of children with maternal measles antibody | 20 weeks of age
  Children with maternal measles antibody
Proportion of children with maternal measles antibody | 9 months of age
  Children with maternal measles antibody
Yellow fever viral load after yellow fever vaccine | 9 months of age
  The level of yellow fever virus in the blood following yellow fever vaccine

SECONDARY OUTCOMES:
Measles antibody levels in the women | 4 weeks after MV or BCG vaccine
  Measles antibody levels in the women
Measles antibody levels in children | 13.5 months of age
  Measles antibody levels in the children
Incidence of morbidity in women after MV or BCG compared with placebo | Up to 12 months following vaccination
  Diseases occurring post-randomisation in women
Incidence of morbidity in children subsequently born to BCG, MV or placebo vaccinated mothers | Up to age 13.5 months
  Diseases occurring in children of randomised women

CONTACTS AND LOCATIONS:
Overall Officials: Christine Benn, DMSc, Principal Investigator — University of Southern Denmark
Locations (1):
- Bandim Health Project, Bissau, Bissau Codex, Guinea-Bissau

IPD SHARING:
Plan to Share IPD: No
The data collected is strictly confidential health data